CLINICAL TRIAL: NCT06010121
Title: Comparison of Bioavailability of Liposomal and Traditional Formulation of Vitamin D3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 02-AP-VD
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Bioavailability of Vitamin D
Keywords: Liposovit-D; Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Vitamin D (Experimental): Daily oral dose of liposomal vitamin D for 4 weeks
  Interventions: Dietary Supplement: Liposomal Vitamin D
- Traditional Vitamin D (Active Comparator): Daily oral dose of traditional vitamin D for 4 weeks
  Interventions: Dietary Supplement: Traditional Vitamin D

INTERVENTIONS:
Dietary Supplement: Liposomal Vitamin D — 2000 IU of cholecalciferol in liposomal formulation
  Arms: Liposomal Vitamin D
Dietary Supplement: Traditional Vitamin D — 2000 IU of cholecalciferol in traditional formulation
  Arms: Traditional Vitamin D

SUMMARY:
The aim of the study was to compare the profiles of 25-hydroxyvitamin D serum concentration in healthy adults after 4 weeks of using vitamin D supplementation either in a liposomal or a traditional formulation.

DETAILED DESCRIPTION:
The study will be randomized, cross-over, participants will be randomly assigned to one of the study groups: A) the group receiving vitamin D3 in traditional formulation B) the group receiving vitamin D3 in liposomal formulation. The day before the start of supplementation (T0), 2 weeks (T1) and 4 weeks (T2) after the start of supplementation, participants will have their blood drawn. Then, after a wash-out period of 2 months, the groups will be switched. Participants will again receive daily supplementation with vitamin D3 for 4 weeks. Blood will be drawn before the start of supplementation (T0), 2 weeks (T1) and 4 weeks (T2) after the start of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18-60 years old.
* Signed informed consent.
* No injuries or hospitalizations within the last 3 months.
* No vitamin D supplementation for the 2 months prior to the study initiation.
* Refraining for the period of the clinical trial from consuming foods additionally fortified with vitamin D and dietary supplements containing vitamin D
* Refraining for the period of the clinical trial from the use of cosmetic therapies that use prolonged body illumination

Exclusion Criteria:

* Unwilling to give consent
* Injuries within the last 3 months
* Obesity, BMI above 30
* Bariatric surgery
* Cystic fibrosis, celiac disease, Crohn's disease
* Metabolic diseases
* Drugs reducing cholesterol absorption, thiazide diuretics, glucocorticosteroids, anticonvulsants, calcium-containing preparations,
* Planned prolonged exposure to sunlight during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Level of 25-hydroxycholecalciferol | Baseline, 2 weeks, 4 weeks
  Comparison of the level of 25(OH)D3 achieved in the blood

CONTACTS AND LOCATIONS:
Locations (1):
- Gdański Uniwersytet Medyczny, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No